CLINICAL TRIAL: NCT02585102
Title: Increasing the Relative Reinforcing Values of Vegetables by Incentive Sensitization
Brief Title: Motivating Value of Vegetables Study
Acronym: VegUp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: USDA, Western Human Nutrition Research Center (U.S. Federal Agency); University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GFHNRC099
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Overweight; Obesity
Keywords: Vegetables
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recommended Vegetables (Other): Diet provided consisting of recommended vegetable intake per Dietary Guidelines for Americans amounts for 8 weeks.
  Interventions: Other: Recommended Vegetable Intake
- Usual Vegetables (Other): Diet consisting of usual vegetable intake amounts for 8 weeks.
  Interventions: Other: Usual Vegetable Intake

INTERVENTIONS:
Other: Recommended Vegetable Intake — Subjects will consume vegetables in amounts recommended by the Dietary Guidelines for Americans
  Arms: Recommended Vegetables
Other: Usual Vegetable Intake — Subjects will consume vegetables in their usual amount
  Arms: Usual Vegetables

SUMMARY:
The purpose of this study is to see if perceived barriers to vegetable consumption can be overcome by making it easier for people eat more vegetables and to see if the effects last over time.

DETAILED DESCRIPTION:
High vegetable consumption is associated with maintenance of a healthy body weight. Americans do not eat vegetables in the amounts recommended by the dietary guidelines and interventions to increase intake have had limited results. Reported barriers to consumption include not knowing how to prepare them and being unused to eating them.To get people to eat vegetables, they have to be motivated to do so. Repeated consumption of snack foods increases overweight and obese individuals' motivation to eat snack foods. The investigators hypothesize that by increasing people's consumption of vegetables by making them easy to eat will increase the motivation value of vegetables. For this study the investigators propose to provide minimally-processed (cleaned, packaged) vegetables to overweight and obese individuals. The motivating value of vegetables will be measured using a computer task where people play a game to earn points towards portions of a vegetable or a neutral food (crackers). The investigators will determine potential moderators of the increase in the motivating value of vegetables such as genetics (single nucleotide polymorphisms) that are associated with the motivating value of food and whether people substitute eating vegetables for other foods. The investigators will also determine changes in adiposity as a result of vegetable consumption. Lastly, the investigators will determine if repeated consumption increases psychosocial predictors of vegetable intake, such as self-efficacy of eating vegetables.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 kg/m2
* Currently eating ≤ 1 cup of vegetables (apart from fried potatoes) per day
* Willing to consent to study conditions

Exclusion Criteria:

* BMI < 25 kg/m2
* Age < 18 years or > 65 years
* Currently dieting or following specific diet
* Allergies or unwillingness to consume study foods
* Gastrointestinal disorder or disease
* Pregnant, lactating, or planning pregnancy
* Current smoker or tobacco user
* High dietary restraint or certain eating patterns
* Inability to give consent
* Medications that would influence appetite, weight gain, or weight loss
* Exclusionary medications: Didrex, Tenuate, Belviq, Contrave, Phendimetrazine, Adipex-P, Suprenza, Xenical, Qsymia, Saxenda

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Change in relative reinforcing value (RRV) of vegetables as assessed by indicator | 0, 4, 8, 12, 16 weeks
  RRV of vegetables will be assessed by evaluating the number of responses (mouse button presses) a participant is willing to complete to gain access to a vegetable or an alternative snack food.

SECONDARY OUTCOMES:
Change in happiness in response to eating vegetables | 0, 8 weeks
  Happiness will be assessed using a validated questionnaire, the "4-item Subjective Happiness Scale," a 7 point Likert scale with 1=not a very happy person to 7=a very happy person, before and after consuming Dietary Guidelines for Americans (DGA) recommended amounts of vegetables.

CONTACTS AND LOCATIONS:
Overall Officials: James N Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casperson SL, Jahns L, Duke SE, Nelson AM, Appleton KM, Larson KJ, Roemmich JN. Incorporating the Dietary Guidelines for Americans Vegetable Recommendations into the Diet Alters Dietary Intake Patterns of Other Foods and Improves Diet Quality in Adults with Overweight and Obesity. J Acad Nutr Diet. 2022 Jul;122(7):1345-1354.e1. doi: 10.1016/j.jand.2022.03.008. Epub 2022 Mar 9. PMID 35278698
- [Derived] Cao JJ, Roemmich JN, Sheng X, Jahns L. Increasing Vegetable Intake Decreases Urinary Acidity and Bone Resorption Marker in Overweight and Obese Adults: An 8-Week Randomized Controlled Trial. J Nutr. 2021 Nov 2;151(11):3413-3420. doi: 10.1093/jn/nxab255. PMID 34386816
- [Derived] Casperson SL, Jahns L, Temple JL, Appleton KM, Duke SE, Roemmich JN. Consumption of a Variety of Vegetables to Meet Dietary Guidelines for Americans' Recommendations Does Not Induce Sensitization of Vegetable Reinforcement Among Adults with Overweight and Obesity: A Randomized Controlled Trial. J Nutr. 2021 Jun 1;151(6):1665-1672. doi: 10.1093/jn/nxab049. PMID 33758940